CLINICAL TRIAL: NCT03932487
Title: The Relationship Between Urine Iodine, Urine Bisphenol A and Autoimmune Thyroid Disease in Reproductive Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiaomei Zhang (Other)
Responsible Party: Sponsor-Investigator, Xiaomei Zhang, Director, Head of endocrinology department., Peking University International Hospital
Organization: Peking University International Hospital (Other)
Other Study IDs: Peking UIH
Record Dates: First submitted 2019-04-24; First posted 2019-04-30 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: The Effect of Iodine and BPA on AITD in Reproduction Women
Keywords: iodine; bisphenol A; autoimmune thyroid disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AITD group: Thyroid antibody positive and hypothyroidism
  Interventions: Other: urinary iodine and urine BPA
- normal group: Thyroid antibody negative and hypothyroidism
  Interventions: Other: urinary iodine and urine BPA

INTERVENTIONS:
Other: urinary iodine and urine BPA — urinary iodine and urine BPA

SUMMARY:
Autoimmune thyroid disease (AITD) is the main cause of hypothyroidism in reproduction women, iodine and bisphenol A are the environmental factors for AITD. The research was mainly designed to investigate the effect of iodine and BPA on AITD in reproduction women to provide new evidence for hypothyroidism in reproduction women.

DETAILED DESCRIPTION:
71 patients with thyroid autoantibody positive were treated as AITD group, another 71 healthy reproduction women were selected as normal group. Women age, BMI, thyroid disease history, family history, marital and reproductive history, whether the application of iodized salt, thyroid function and thyroid autoantibodies detection were recorded. Meanwhile urine iodine, urinary iodine/urinary creatinine, urine BPA and urinary BPA/creatinine were tested. The urine iodine and BPA levels of the two groups were compared. Taking AITD as the dependent variable, logistic regression was conducted to analyze whether urinary iodine and BPA were risk factors of AITD.

ELIGIBILITY:
Inclusion Criteria:

1. AITD group: positive thyroid autoantibody (one thyroid autoantibody), normal thyroid function.
2. Normal group: thyroid autoantibody negative, normal thyroid function.
3. No previous history of hyperthyroidism or hypothyroidism, no history of thyroid surgery or I131 radiotherapy, and no thyroid hormone or anti-thyroid drugs were used.

Exclusion Criteria:

1. Patients with severe liver, kidney, heart and other important organ failure.
2. Merger with other autoimmune diseases.
3. Amiodarone, iodine contrast agent and other drugs affecting thyroid function are used.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In Peking University international hospital women of childbearing age (age 20 to 45 years old) of 142 cases of 71 patients with thyroid autoantibodies positive as AITD group, the other selected 71 cases of healthy women of childbearing age as normal group, record the age, BMI, and examination of the history of history of thyroid disease, family history and whether the application of iodized salt and other general information and we, thyroid autoantibodies detection results, urine iodine, urinary iodine/urinary creatinine and urinary BPA and urinary BPA/creatinine detection.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Estimated)
Dates: Start 2019-06-24 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of urinary iodine levels between the two groups | 2019-2011
  Urinary iodine levels were compared between patients with autoimmune thyroid disease and normal women.
Comparison of urinary BPA levels between the two groups | 2019-2011
  Urinary BPA levels were compared between patients with autoimmune thyroid disease and normal women.

SECONDARY OUTCOMES:
Influencing factors of autoimmune thyroid diseases. | 2019-2012
  Abnormal levels of iodine and PBA are influential factors in autoimmune thyroid disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University international hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Urinary iodine and bisphenol A may affect AITD in reproduction women.